CLINICAL TRIAL: NCT02223169
Title: Dietary Intervention Study to Assess the Effects of Albumin-Derived Peptides on Cardio-Metabolic Risk Factors in Adults
Brief Title: Human Intervention Study of Egg Protein Derivative on Cardiovascular Risk
Acronym: CardiProtein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Mairead Kiely PhD, Dr, University College Cork
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ECFP7-312090
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Blood Pressure; Hypertension; Cardiovascular disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Egg albumin-derived peptide (Experimental): Each participant will consume 1 sachet of Egg albumin-derived peptide (3 g) each day mixed with a fruit juice drink for 42 days.
  Interventions: Dietary Supplement: Egg albumin-derived peptide
- Placebo (Placebo Comparator): Participants will consume one sachet of the placebo mixed with a fruit juice drink that will appear and taste similar to the albumin derived peptide sachet.
  Interventions: Dietary Supplement: Egg albumin-derived peptide

INTERVENTIONS:
Dietary Supplement: Egg albumin-derived peptide — Double-blind intervention study cross-over design with one sachet containing 3g Egg albumin-derived peptide (Tensio-control) or placebo (maltodextrin) in Phase one followed by cross-over in Phase 2.
  Other Names: Tensio-control

SUMMARY:
Heart disease and stroke are the most common cause of death in Ireland today.One of the main risk factors for heart disease and stroke is high blood pressure or hypertension. Research has found that certain specific proteins or peptides found in foods such as dairy, meat, fish and eggs may promote heart health reducing blood pressure in adults with hypertension. The aim of this study is to investigate the potential beneficial effects egg peptides may have on heart health, in particular, effects on blood pressure.

DETAILED DESCRIPTION:
Poor dietary habits of Irish adults has been accompanied by epidemics of obesity and metabolic disorders such as type II diabetes leading to a substantial predicted increase in the prevalence of chronic diseases such as cardiovascular disease.Hypertension is a major contributing factor to the development of cardiovascular and metabolic diseases. Dietary factors play a significant role in the prevention and/or treatment of hypertension and therefore the development of foods with antihypertensive properties could prove beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Non-diabetic
* Aged 50-65
* BMI 25-35kg/m²
* Mild hypertensive: Blood pressure 130-149 mmHg

Exclusion Criteria:

* Current smoker
* Diagnosed hypertensive
* History of cardiovascular disease
* Diabetic
* Chronic kidney disease
* Gastrointestinal disease
* Currently on anti-hypertensive medications
* Allergic to eggs

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
A change between baseline blood pressure and endpoint blood pressure within the intervention group vs control group. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Mairead Kiely, PhD, Principal Investigator — University College Cork
Locations (2):
- Ireland (2):
  - School of Food and Nutritional Sciences, UCC, Cork
  - University College Cork, Cork